CLINICAL TRIAL: NCT04309214
Title: Market Research - Acceptability Study for a Range of New MCT Based Products (Dr Schär - Kanso) Kanso DeliMCT 53% (Cream) Kanso DeliMCT 28% (Tomato or Mushroom) Kanso DeliMCT 21% (Cacaobar)
Brief Title: Market Research - Acceptability Study for New MCT Fat Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Schär AG / SPA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Kanso 2
Record Dates: First submitted 2020-03-09; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Ketosis; Epilepsy; Fatty Acid Oxidation Disorder; Malabsorption; Ketogenic Diet; Medium Chain Triglycerides
MeSH Terms: conditions — Ketosis; Epilepsy; Malabsorption Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MCT fats (Experimental): MCT fats to be consumed, one portion per day to ensure tolerance and compliance to the product whilst support the dietary management for a range if disease states namely, the ketogenic diet, fatty acid oxidation disorders and malabsorption.
  Interventions: Dietary Supplement: MCT fats

INTERVENTIONS:
Dietary Supplement: MCT fats — Subjects will be asked to take 3 new MCT products for 7 days each over a 25 day period
  Other Names: medium chain triglycerides

SUMMARY:
This is a market research, observational study to evaluate the tolerability and acceptability of MCT supplements for young children, young people and adults with intractable epilepsy, GLUT-1 or PDHD from 3 years to adulthood.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epilepsy requiring a ketogenic or a specialist diet as part of their treatment.
* Subjects new to taking or who are already taking an MCT product and are willing to try each of the 3 study products for 7 days each. 21 days taking product with 2 days between each new product trialled.
* Those patients who have been taking MCT in their diet should do so for a minimum of 4 weeks before commencement of the study.
* Patients aged 3 years of age to adulthood.
* Written informed consent obtained from patient or parental caregiver.

Exclusion Criteria:

* Presence of serious concurrent illness
* Investigator's uncertainty about the willingness or ability of the patient to comply with the protocol requirements
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study
* Any patients having taken antibiotics over the previous 2 weeks leading up to the study
* Patients already on and MCT product who have been taking it in their diet for less than 4 weeks
* Patients less than 3 years of age
* Patients over 20 years.

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerance | 7 days for each product, maximum 25 days
  Questionnaire detailing any GI symptoms, severity and change from usual The collection of daily data about the gastrointestinal tolerance of the product
Product compliance | 7 days for each product, maximum 25 days
  Daily questionnaire on amounts offered and amounts actually consumed, compared to recommended amount.
Product palatability | 7 days for each product, maximum 25 days
  Questionnaire data captured to evaluate taste
Product acceptability | 7 days for each product, maximum 25 days
  Brief tick-box questionnaire on overall liking and acceptability of product

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Aberdeen Children's Hospital, Aberdeen, Grampian, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This study will be used for the registration and reimbursement for the products used as foods for special medical purposes.